CLINICAL TRIAL: NCT01243177
Title: A Multicenter, Double-blind, Double-dummy, Randomized, Positive- Controlled Study Comparing the Efficacy and Safety of Lacosamide (200 to 600 mg/Day) to Controlled Release Carbamazepine (400 to 1200 mg/Day), Used as Monotherapy in Subjects (≥ 16 Years) Newly or Recently Diagnosed With Epilepsy and Experiencing Partial-onset or Generalized Tonic-clonic Seizures.
Brief Title: Trial Comparing the Efficacy and Safety of Lacosamide (LCM) to Carbamazepine Controlled-Release (CBZ-CR); Initial Monotherapy in Epilepsy; Subjects Aged 16 and Older
Acronym: SP0993
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Eden Sarl (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0993; 2010-019765-28 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Epilepsy; Monotherapy
Keywords: Lacosamide; Vimpat®; Epilepsy; Monotherapy; Velocity
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lacosamide (Experimental)
  Interventions: Drug: Lacosamide
- Carbamazepine-Controlled Release (CBZ-CR) (Active Comparator)
  Interventions: Drug: Carbamazepine-Controlled Release

INTERVENTIONS:
Drug: Lacosamide — Lacosamide:
  * Strengths: 50 mg / 100 mg
  * Form: tablets
  * Dosage: total daily target dose of 200 mg, 400 mg or 600 mg. 1 dose reduction was allowed from either 600 mg to 500 mg or from 400 mg to 300 mg total daily dose
  * Duration: up to 118 weeks
  Other Names: Vimpat®
  Arms: Lacosamide
Drug: Carbamazepine-Controlled Release — Carbamazepine-CR:
  * Strengths: 200 mg
  * Form: tablets
  * Dosage: total daily target dose of 400 mg, 800 mg or 1200 mg. 1 dose reduction was allowed from either 1200 mg to 1000 mg or from 800 mg to 600 mg total daily dose
  * Duration: up to 118 weeks
  Other Names: Tegretol® Retard Tablets 200 mg
  Arms: Carbamazepine-Controlled Release (CBZ-CR)

SUMMARY:
Compare efficacy and safety of Lacosamide (LCM) to Carbamazepine Controlled-Release (CBZ-CR) as monotherapy in newly or recently newly diagnosed subjects with a primary efficacy endpoint of 6-month seizure freedom. Noninferiority design to show a similar risk/benefit balance between Lacosamide (LCM) and Carbamazepine-CR (CBZ-CR).

ELIGIBILITY:
Inclusion Criteria:

* Subject able to comply with study requirements
* Subject is 16 years and older (female; male). Minors will be included in countries only if legally permitted
* Subject has newly or recently diagnosed Epilepsy experiencing partial onset seizures (POS) or generalized tonic-clonic seizures with at least 2 unprovoked seizures separated by 48 hours in the 12 months preceding Visit 1 out of which at least 1 seizure occured 3 months preceding Visit 1
* Subject has had an Electroencephalogram (EEG) and a brain Computed Tomography (CT) scan or Magnetic Resonance Imaging (MRI) exam of the brain within the past 12 months. If the EEG and brain CT scan or MRI exam were not performed prior to Visit 1, they need to be completed and results must be available prior to randomization at Visit 2

Exclusion Criteria:

* Subject has a history or presence of seizures of other types than partial-onset (IA, IB, IC with clear focal origin) and generalized tonic-clonic (without clear focal origin) seizures (eg, myoclonic, absence)
* Subject has a history or presence of seizures occurring only in clustered patterns, defined as repeated seizures occurring over a short period of time (ie, < 20 minutes) with or without function regained between 2 ictal events
* Subject has a history, clinical, or Electroencephalogram (EEG) finding suggestive of Idiopathic Generalized Epilepsy (IGE) at randomization
* Subject has current or previous diagnosis of pseudoseizures, conversion disorders, or other nonepileptic ictal events that could be confused with seizures based on expert opinion and/or EEG evidence
* Subject has any medical or psychiatric condition
* Subject has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response (Yes) to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening
* Subject has received treatment with Phenobarbital or Primidone within 28 days prior to Visit 1
* Subject is taking Benzodiazepines for a nonepilepsy indication
* Subject has been treated for Epilepsy with any Antiepileptic Drug (AED) (including Benzodiazepines) in the last 6 months before Visit. However, acute and subacute seizure treatment is accepted with a maximum of 2 weeks duration and if treatment was stopped at least 3 days prior to randomization
* Prior use of Felbamate or Vigabatrin is not allowed
* Benzodiazepines as rescue therapy for Epilepsy may have been used as needed in this time period, but not more frequently than once per week
* Subject has a medical condition that could reasonably be expected to interfere with drug absorption, distribution, metabolism, or excretion, has a history of alcohol or drug abuse within the previous 2 years
* Asian ancestry and tests positive for HLA-B*1502 allele
* Asian ancestry and tests positive for HLA-A*3101 allele

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 888 (Actual)
Dates: Start 2011-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (184):
- United States (15):
  - 786, Alabaster, Alabama
  - 799, Huntsville, Alabama
  - 780, Phoenix, Arizona
  - 777, Little Rock, Arkansas
  - 795, Ocala, Florida
  - 789, Panama City, Florida
  - 776, Port Charlotte, Florida
  - 779, Manhattan, Kansas
  - 874, Charlotte, North Carolina
  - 876, Hickory, North Carolina
  - 873, Raleigh, North Carolina
  - 794, Oklahoma City, Oklahoma
  - 881, Mansfield, Texas
  - 790, Madison, Wisconsin
  - 798, Casper, Wyoming
- Australia (9):
  - 106, East Gosford, New South Wales
  - 109, Randwick, New South Wales
  - 102, Westmead, New South Wales
  - 103, Herston, Queensland
  - 100, Woodville, South Australia
  - 101, Fitzroy, Victoria
  - 108, Heidelberg, Victoria
  - 104, Chatswood
  - 105, Clayton
- Belgium (4):
  - 127, Bruges
  - 134, Bruges
  - 128, Hasselt
  - 126, Leuven
- Bulgaria (8):
  - 805, Blagoevgrad
  - 807, Panagyurishte
  - 803, Pleven
  - 810, Rousse
  - 806, Sofia
  - 808, Sofia
  - 811, Sofia
  - 809, Veliko Tarnovo
- Canada (6):
  - 153, St. John's, Newfoundland and Labrador
  - 152, Greenfield Park, Quebec
  - 155, Calgary
  - 158, Halifax Nova Scotia
  - 156, Hamilton
  - 159, Veilleux
- Czechia (5):
  - 185, Brno
  - 190, Ostrava - Vitkovice
  - 184, Prague
  - 189, Prague
  - 180, Zlín
- Finland (2):
  - 205, Helsinki
  - 207, Kuopio
- France (4):
  - 236, Nancy
  - 233, Paris
  - 231, Strasbourg
  - 235, Toulouse
- Germany (13):
  - 263, Altenburg
  - 258, Aschaffenburg
  - 265, Bad Neustadt an der Saale
  - 257, Berlin
  - 262, Berlin
  - 270, Berlin
  - 271, Cologne
  - 260, Göttingen
  - 269, Leipzig
  - 256, Marburg
  - 264, München
  - 261, Münster
  - 259, Osnabrück
- Greece (4):
  - 496, Alexandroupoli
  - 495, Ioannina
  - 493, Thessaloniki
  - 490, Thessalonikis
- Hungary (9):
  - 289, Balassagyarmat
  - 283, Budapest
  - 284, Budapest
  - 286, Debrecen
  - 282, Győr
  - 288, Pécs
  - 285, Szeged
  - 290, Szekszárd
  - 291, Szombathely
- Italy (5):
  - 310, Bari
  - 309, Modena
  - 308, Padua
  - 314, Prato
  - 311, Roma
- Japan (14):
  - 831, Asaka-shi
  - 833, Hamamatsu
  - 834, Kagoshima
  - 844, Kamakura-shi
  - 846, Kawasaki-shi
  - 829, Kokubunji-shi
  - 843, Miyakonojō
  - 835, Nagoya
  - 830, Nara
  - 837, Okayama
  - 828, Saitama-shi
  - 836, Sapporo
  - 847, Sapporo
  - 832, Shizuoka
- 751, Riga, Latvia
- Lithuania (3):
  - 727, Alytus
  - 724, Kaunas
  - 728, Vilnius
- 547, San Luis Potosí City, Mexico
- Philippines (3):
  - 673, Manila
  - 672, Pasig
  - 676, Quezon City
- Poland (7):
  - 336, Gdansk
  - 334, Katowice
  - 340, Katowice
  - 342, Lublin
  - 341, Poznan
  - 338, Szczecin
  - 343, Warsaw
- Portugal (5):
  - 360, Coimbra
  - 362, Lisbon
  - 365, Lisbon
  - 366, Porto
  - 361, Santa Maria da Feira
- Romania (8):
  - 576, Bucharest
  - 569, Cluj-Napoca
  - 578, Craiova
  - 570, Iași
  - 579, Iași
  - 571, Sibiu
  - 577, Sibiu
  - 572, Târgu Mureş
- Russia (11):
  - 387, Kazan'
  - 389, Kazan'
  - 396, Kirov
  - 394, Moscow
  - 401, Moscow
  - 390, Nizhny Novgorod
  - 392, Novosibirsk
  - 397, Saint Petersburg
  - 400, Saint Petersburg
  - 386, Smolensk
  - 399, Yaroslavl
- Slovakia (7):
  - 594, Dolný Kubín
  - 598, Dubnica nad Váhom
  - 596, Hlohovec
  - 600, Krompachy
  - 595, Levoča
  - 599, Tornaľa
  - 601, Žilina
- South Korea (9):
  - 525, Busan
  - 521, Daegu
  - 518, Dajeon
  - 516, Seoul
  - 517, Seoul
  - 519, Seoul
  - 520, Seoul
  - 523, Seoul
  - 524, Seoul
- Spain (10):
  - 422, Badalona
  - 413, Barcelona
  - 418, Donostia / San Sebastian
  - 416, Madrid
  - 425, Madrid
  - 426, Madrid
  - 421, Murcia (El Palmar)
  - 419, San Cristóbal de La Laguna
  - 414, Santiago de Compostela
  - 424, Seville
- Sweden (3):
  - 440, Gothenburg
  - 438, Stockholm
  - 442, Umeå
- Switzerland (4):
  - 651, Aarau
  - 654, Biel
  - 653, Lugano
  - 647, Sankt Gallen
- Thailand (4):
  - 699, Bangkok
  - 702, Bangkok
  - 703, Bangkok
  - 698, Khon Kaen
- Ukraine (7):
  - 622, Chernihiv
  - 628, Dnipropetrovsk
  - 626, Kharkiv
  - 621, Luhansk
  - 625, Odesa
  - 632, Simferopol
  - 633, Vinnytsa
- United Kingdom (3):
  - 466, Birmingham
  - 472, Glasgow
  - 471, Stoke-on-Trent

REFERENCES:
- [Result] Baulac M, Rosenow F, Toledo M, Terada K, Li T, De Backer M, Werhahn KJ, Brock M. Efficacy, safety, and tolerability of lacosamide monotherapy versus controlled-release carbamazepine in patients with newly diagnosed epilepsy: a phase 3, randomised, double-blind, non-inferiority trial. Lancet Neurol. 2017 Jan;16(1):43-54. doi: 10.1016/S1474-4422(16)30292-7. Epub 2016 Nov 24. PMID 27889312
- [Result] Mintzer S, Dimova S, Zhang Y, Steiniger-Brach B, De Backer M, Chellun D, Roebling R. Effects of lacosamide and carbamazepine on lipids in a randomized trial. Epilepsia. 2020 Dec;61(12):2696-2704. doi: 10.1111/epi.16745. Epub 2020 Nov 17. PMID 33200428
- [Derived] Lindauer A, Laveille C, Stockis A. Time-to-Seizure Modeling of Lacosamide Used in Monotherapy in Patients with Newly Diagnosed Epilepsy. Clin Pharmacokinet. 2017 Nov;56(11):1403-1413. doi: 10.1007/s40262-017-0530-8. PMID 28290119
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll in April 2011 and concluded in August 2015.
Pre-assignment Details: Participant Flow refers to the Safety Analysis Set which is defined as all randomized subjects who took at least 1 dose of study medication and is identical with the Full Analysis Set.
Groups:
- Lacosamide: * Strengths: 50 mg / 100 mg
  * Form: tablets
  * Dosage: total daily target dose of 200 mg, 400 mg or 600 mg. 1 dose reduction was allowed from either 600 mg to 500 mg or from 400 mg to 300 mg total daily dose
  * Duration: up to 118 weeks
- Carbamazepine-Controlled Release (CBZ-CR): * Strengths: 200 mg
  * Form: tablets
  * Dosage: total daily target dose of 400 mg, 800 mg or 1200 mg. 1 dose reduction was allowed from either 1200 mg to 1000 mg or from 800 mg to 600 mg total daily dose
  * Duration: up to 118 weeks
Period: Overall Study
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Started | 444 | 442
Completed | 266 | 264
Not Completed | 178 | 178
Not completed — Lack of Efficacy | 47 | 31
Not completed — Protocol Violation | 11 | 10
Not completed — Lost to Follow-up | 15 | 18
Not completed — Withdrawal by Subject | 46 | 38
Not completed — AE, serious fatal | 0 | 1
Not completed — SAE, non-fatal | 7 | 9
Not completed — AE, non-serious non-fatal | 40 | 58
Not completed — SAE, fatal + SAE, non-fatal | 1 | 0
Not completed — SAE,non-fatal+AE,non-serious non-fatal | 0 | 1
Not completed — Other Reason | 11 | 12

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Analysis Set which is defined as all randomized subjects who took at least 1 dose of study medication and is identical with the Full Analysis Set.
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR) | Total Title
Number analyzed (Participants) | 444 | 442 | 886
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 19 | 46
  Between 18 and 65 years | 355 | 366 | 721
  >=65 years | 62 | 57 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (17.9) | 41.8 (17.2) | 41.8 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 210 | 411
  Male | 243 | 232 | 475

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in the Full Analysis Set (FAS) Remaining Seizure Free for 6 Consecutive Months (26 Consecutive Weeks) of Treatment Following Stabilization at the Last Evaluated Dose for Each Subject
Description: The proportion of subjects remaining seizure free for 6 months (26 weeks) was estimated using Kaplan-Meier methods.
Time Frame: 6 consecutive months (26 consecutive weeks) of treatment following stabilization at the last evaluated dose for each subject
Population: Full Analysis Set (FAS), consisting of all randomized subjects who took at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 444 | 442
percentage of subjects | 89.8 [86.8 to 92.8] | 91.1 [88.2 to 94.0]
Statistical Analysis 1: Comparison: Lacosamide vs Carbamazepine-Controlled Release (CBZ-CR); This was a noninferiority assessment of Lacosamide versus Carbamazepine-CR for the proportion of subjects remaining seizure free for 6 months at the last evaluated dose; Test type: Non-Inferiority or Equivalence — The hypothesis was as follows: H0: [S(t)LCM] - [S(t)CBZ-CR] ≤ -12 % versus HA: [S(t)LCM] - [S(t)CBZ-CR] > -12 %, where S(t) (t= 182 days) is the cumulative rate of subjects remaining seizure free for 6 months following stabilization at the last evaluated dose (also known as the survivorship function), and -12 % represents the noninferiority margin based on absolute difference; Mantel Haenszel; The analysis was stratified based on the number of seizures in the 3 months preceding enrollment (≤ 2 and >2); Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-5.5 to 2.8] — The lower limit of the confidence interval was >-12 %, noninferiority of LCM to CBZ-CR was demonstrated. Additionally, the lower confidence limit relative to the CBZ-CR seizure freedom rate was >- 20 %

2. Primary Outcome: Proportion of Subjects in the Per Protocol Set (PPS) Remaining Seizure Free for 6 Consecutive Months (26 Consecutive Weeks) of Treatment Following Stabilization at the Last Evaluated Dose for Each Subject
Description: The proportion of subjects remaining seizure free for 6 months (26 weeks) was estimated using Kaplan-Meier methods.
Time Frame: 6 consecutive months (26 consecutive weeks) of treatment
Population: The Per Protocol Set (PPS) was defined as containing all subjects in the Full Analysis Set (FAS) who did not have any important protocol deviations determined to impact the interpretation of primary efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 408 | 397
percentage of subjects | 91.4 [88.5 to 94.3] | 92.8 [90.1 to 95.6]
Statistical Analysis 1: Comparison: Lacosamide vs Carbamazepine-Controlled Release (CBZ-CR); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mantel Haenszel; The analysis was stratified based on the number of seizures in the 3 months preceding enrollment (≤ 2 and >2); Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-5.3 to 2.7] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Number of Subjects With at Least One Treatment-emergent Adverse Event (AE) During the Treatment Phase (up to 113 Weeks)
Description: An Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent AEs were defined as AEs that started on or after the date of first dose of study medication and within 30 days following the date of final study medication administration, or AEs whose intensity worsened on or after the date of first dose of study medication and within 30 days following the date of last dose.
Time Frame: Duration of the Treatment Phase (up to 113 weeks)
Population: Safety Analysis Set consisting of all randomized subjects who took at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 444 | 442
Participants | 328 | 332

4. Primary Outcome: Number of Subjects Who Withdraw From the Study Due to a Treatment-emergent Adverse Event (AE) During the Treatment Phase (up to 113 Weeks)
Description: as for outcome 3
Time Frame: Duration of the Treatment Phase (up to 113 weeks)
Population: Safety Analysis Set consisting of all randomized subjects who took at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 444 | 442
Participants | 47 | 69

5. Secondary Outcome: Proportion of Subjects Remaining Seizure Free for 12 Consecutive Months (52 Consecutive Weeks) Following Stabilization at the Last Evaluated Dose for Each Subject
Description: The proportion of subjects remaining seizure free for 12 months (52 weeks) was estimated using Kaplan-Meier methods.
Time Frame: 12 consecutive months of treatment following stabilization at the last evaluated dose for each subject
Population: Full Analysis Set (FAS), consisting of all randomized subjects who took at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 444 | 442
percentage of subjects | 77.8 [73.4 to 82.2] | 82.7 [78.5 to 86.8]

6. Primary Outcome: Number of Subjects With at Least One Treatment-emergent Serious Adverse Event (SAE) During the Treatment Phase (up to 113 Weeks)
Description: An Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  A Serious Adverse Event must meet 1 or more predefined criteria like death, life-threatening, etc. Treatment-emergent AEs were defined as AEs that started on or after the date of first dose of study medication and within 30 days following the date of final study medication administration, or AEs whose intensity worsened on or after the date of first dose of study medication and within 30 days following the date of last dose.
Time Frame: Duration of the Treatment Phase (up to 113 weeks)
Population: Safety Analysis Set consisting of all randomized subjects who took at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 444 | 442
Participants | 32 | 43

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the whole study from Screening Phase (Week 0) over Evaluation, Maintenance and End of Study Phase up to 121 weeks.
Description: Adverse Events refer to the Safety Analysis Set consisting of all randomized subjects who took at least 1 dose of study medication.
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Serious Adverse Events (participants affected / at risk) | 36/444 | 46/442
Other Adverse Events (participants affected / at risk) | 165/444 | 181/442
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=444) | Carbamazepine-Controlled Release (CBZ-CR) (N=442)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Smear cervix abnormal (Investigations) | 1 (1) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 4 (4) | 2 (3)
Complex partial seizures (Nervous system disorders) | 2 (2) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Motor neurone disease (Nervous system disorders) | 1 (1) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Preictal state (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=444) | Carbamazepine-Controlled Release (CBZ-CR) (N=442)
Nausea (Gastrointestinal disorders) | 26 (32) | 23 (30)
Fatigue (General disorders) | 34 (38) | 49 (55)
Nasopharyngitis (Infections and infestations) | 29 (42) | 29 (37)
Gamma-glutamyltransferase increased (Investigations) | 7 (8) | 35 (36)
Headache (Nervous system disorders) | 60 (82) | 58 (78)
Dizziness (Nervous system disorders) | 53 (61) | 41 (52)
Somnolence (Nervous system disorders) | 27 (28) | 41 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days